CLINICAL TRIAL: NCT05029128
Title: Enhancing Skeletal Adaptation to Exercise by Attenuating the Acute Disruption of Calcium Homeostasis During Exercise
Brief Title: Enhancing Skeletal Adaptations to PTH and Exercise
Acronym: ESkAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ENDB-007-20F; 1 I01 CX00284 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2021-08-12; First posted 2021-08-31 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Exercise; Bone Resorption; Bone Formation
Keywords: Acute exercise; Exercise training; Bone resorption; Bone formation; Parathyroid hormone; Calcium homeostasis
MeSH Terms: conditions — Motor Activity; Bone Resorption

STUDY DESIGN:
Intervention Model Description: All participants will undergo the same exercise intervention for this proof-of-concept project, so there is no randomization. The exercise will be treadmill walking at 70-80% of HRmax for 60 min/d, 4 d/wk, for 4 wk. The mode and intensity of exercise were selected because high-intensity weight-bearing exercise is recommended for bone health, and walking is the most common weight-bearing activity. Although "high-intensity" exercise for bone health refers to the intensity of bone-loading forces, %HRmax is a good proxy because peak bone-loading forces increase as walking or running speed increases. Exercise sessions will be supervised by the research team.
  This exercise prescription was used in the studies of young and older adults that provided the scientific premise for the current study and resulted in robust PTH and CTX responses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise (Other): All participants engage in exercise training
  Interventions: Behavioral: Endurance exercise intervention

INTERVENTIONS:
Behavioral: Endurance exercise intervention — All participants engage in treadmill walking 4 days/week, 60 minutes/day, at 70-80% of HRmax for 4 weeks.

SUMMARY:
Exercise is essential for building and maintaining bone mass and strength, but current exercise recommendations for how to achieve this lack detail on the optimal exercise prescription. Recent studies found that blood calcium level decreases during exercise, and that calcium is mobilized from bone to slow the decline. If this occurs repeatedly during exercise training, it could diminish the potential benefits of exercise to improve bone health. The proposed study will determine whether further research on pre-exercise supplemental calcium to minimize the decline in blood calcium level during exercise is warranted. This research is important for Veterans because they are at increased risk of hip fracture when compared with non-Veterans. Further, because osteoporosis in men is under-recognized and under-treated, providing male (and female) Veterans with more specific exercise and nutrition guidelines has the potential to enhance bone health, reduce fracture risk, and improve quality of life.

DETAILED DESCRIPTION:
Exercise is essential for building and maintaining bone mass and strength, but recent work has raised the possibility that current exercise recommendations for bone health may not be appropriate. There is strong evidence that a single bout of vigorous exercise has an acute catabolic effect in bone (i.e., increased resorption) that lasts several hours. This is mediated by a decrease in serum calcium (Ca) during exercise, which stimulates parathyroid hormone (PTH) secretion. PTH then activates bone resorption to mobilize Ca from bone, presumably to prevent the decrease in serum Ca from progressing to a harmful level. This cascade of events can be markedly attenuated by minimizing the decline in serum Ca during exercise via either intravenous or oral Ca administration. The timing of Ca supplementation relative to exercise is likely important, because it must be available for gut absorption during exercise. Interestingly, repeated pharmacologic stimulation of the PTH receptor with PTH analogs (teriparatide, abaloparatide) has anabolic effects on bone, suggesting that repeated exercise-induced increases in PTH could have a chronic anabolic skeletal effect, in addition to the acute catabolic effect, which may be apparent only after repeated exercise sessions. If this is the case, suppressing the PTH response with pre-exercise Ca supplementation may not be appropriate. In this context, this proof-of-concept study will include a short exercise intervention consisting of treadmill exercise at 70% to 80% of maximal heart rate, 60 minutes per day, 4 days per week, for 4 weeks. Serum markers of bone formation and resorption will be measured before, during, and for 24 hours after the 1st, 8th, and 16th exercise sessions to address two questions: 1) Does the acute catabolic response of bone to a single bout of exercise continue to occur with repeated exercise sessions (i.e., exercise training)? 2) Does exercise training also generate an anabolic PTH-mediated bone response, similar to the anabolic response to PTH analog therapy? If the answers to questions 1 and 2 are YES (persistent catabolic signal) and NO (lack of anabolic signal), this will support the need for the randomized controlled trial (RCT), which will evaluate whether taking Ca before exercise to attenuate the acute catabolic response improves skeletal adaptations to exercise training. The overarching goal is to improve the currently imprecise recommendations for exercise to improve and maintain bone health. This research is of high relevance to Veterans, who are at increased risk of hip fracture when compared with non-Veterans. Further, because osteoporosis in men is under-recognized, under-diagnosed, and under-treated, providing male Veterans with an effective non-pharmacologic therapeutic option to reduce fracture risk may help close this treatment gap. The potential impact of this research also extends beyond Veterans. It could lead to reduced risk of exercise-related bone injury (i.e., stress fractures) in active duty military personnel and athletes and to improved bone health in the general population.

ELIGIBILITY:
Inclusion Criteria:

Female and male Veterans aged 25 to 45 y and 55 to 75 y will be enrolled. Eligible volunteers will be normally active (e.g., recreational cycling or walking) but will not participate in regular moderate-to-vigorous exercise. Women will be premenopausal with regular menstrual cycles or postmenopausal, defined as absence of menses for at least 12 mo or, in those who underwent a hysterectomy, a serum follicle stimulating hormone (FSH) >30 mIU/mL.

Exclusion Criteria:

* Initiation or change in dose in the past 6 months of medications that affect bone metabolism

  * e.g., osteoporosis medications, thiazide/loop diuretics, systemic glucocorticoids
* BMD T-score <-2.5 at the total hip, femoral neck, or lumbar spine
* Impaired renal function, defined as an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2
* Abnormal alkaline phosphatase
* Untreated thyroid dysfunction, defined as an ultrasensitive thyroid stimulating hormone (TSH) <0.5 or >5.0 mU/L
* Serum Ca <8.5 or >10.3 mg/dL
* Serum 25(OH)D <20 ng/mL
* Uncontrolled hypertension (resting systolic blood pressure (BP) >150 mmHg or diastolic BP >90 mmHg)
* Type 1 diabetes
* Type 2 diabetes if on insulin or sulfonylurea therapy
* hemoglobin A1c >7%
* Cardiovascular disease; defined as subjective or objective indicators of ischemic heart disease (e.g., angina, ST segment depression) or serious arrhythmias at rest or during the graded exercise test (GXT)

  * volunteers who have a positive GXT can be re-considered after follow-up evaluation by a cardiologist
* Anemia (hemoglobin <12.1 g/dL for women, <14.3 g/dL for men)
* Fracture in the past 6 months
* Body mass index >39 kg/m2

  * In the event of abnormal eGFR, alkaline phosphatase, TSH, BP, 25(OH)D, or hemoglobin values, volunteers can be reassessed, including after appropriate follow-up evaluation and treatment by their health care provider

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
C-terminal peptide of type 1 collagen (CTX) | The primary outcome for Aim 1 is the change in CTX (dCTX) from before exercise to the peak during 4 hours of recovery measured during the 1st, 8th, and 16th exercise sessions.
  CTX is a marker of bone resorption. An increase in CTX in response to exercise is evidence of an acute catabolic response of bone.
Procollagen 1 intact N-terminal propeptide (P1NP) | The primary outcome for Aim 2 is the change in the pre-exercise P1NP (15 minutes before the start of exercise) from the 1st to the 16th exercise session.
  P1NP is a marker of bone formation. An increase in P1NP from before to after an exercise intervention is evidence of an anabolic response of bone.

SECONDARY OUTCOMES:
P1NP | Serum P1NP is measured before (-15, 0 minutes), during (15, 30, 45, 60 minutes), and after (15, 30, 60, 120, 180, 240 minutes, 24 hours) the 1st, 8th, and 16th exercise sessions
  Serum P1NP is measured to determine if there is an acute anabolic response of bone to exercise and whether it changes in response to exercise training
Urinary calcium excretion (uCa) | Urinary Ca excretion is measured over the 4 hours of recovery after the 1st, 8th, and 16th exercise sessions
  Urinary tCa is used to account for Ca loss subsequent to the activation of bone resorption during exercise
Serum ionized Ca (iCa) | Serum iCa is measured before (-15, 0 minutes), during (15, 30, 45, 60 minutes), and after (15, 30, 60, 120, 180, 240 minutes, 24 hours) the 1st, 8th, and 16th exercise sessions
  Serum iCa is measured to assess the stimulus for PTH secretion and to describe the pattern of change in iCa during and after exercise
Serum total Ca (tCa) | Serum tCa is measured before (-15, 0 minutes), during (15, 30, 45, 60 minutes), and after (15, 30, 60, 120, 180, 240 minutes, 24 hours) the 1st, 8th, and 16th exercise sessions
  Serum tCa is measured to help interpret changes in iCa (e.g., changes in Ca binding) and to describe the pattern of change in tCa during and after exercise
Serum parathyroid hormone (PTH) | Serum PTH is measured before (-15, 0 minutes), during (15, 30, 45, 60 minutes), and after (15, 30, 60, 120, 180, 240 minutes, 24 hours) the 1st, 8th, and 16th exercise sessions
  Serum PTH is measured to assess the stimulus for the activation of bone resorption and to describe the pattern of change in PTH during and after exercise
Serum phosphorus (PO4) | Serum PO4 is measured before (-15, 0 minutes), during (15, 30, 45, 60 minutes), and after (15, 30, 60, 120, 180, 240 minutes, 24 hours) the 1st, 8th, and 16th exercise sessions
  Serum PO4 is measured because it is a potential stimulus for PTH secretion
Hematocrit (Hct) | Hct is measured before (-15, 0 minutes), during (15, 30, 45, 60 minutes), and after (15, 30, 60, 120, 180, 240 minutes, 24 hours) the 1st, 8th, and 16th exercise sessions
  Hct is used to adjust iCa, tCa, PTH, CTX, P1NP, and PO4 for the plasma volume contraction that occurs with exercise
Hemoglobin (Hgb) | Hgb is measured before (-15, 0 minutes), during (15, 30, 45, 60 minutes), and after (15, 30, 60, 120, 180, 240 minutes, 24 hours) the 1st, 8th, and 16th exercise sessions
  Hgb is used to adjust iCa, tCa, PTH, CTX, P1NP, and PO4 for the plasma volume contraction that occurs with exercise

OTHER OUTCOMES:
Maximal heart rate (HRmax) | HRmax is measured at baseline during a maximal treadmill test
  HRmax is used to describe the cohort and generate individual exercise prescriptions for the intervention
Peak aerobic power (VO2peak) | VO2peak is measured at baseline during a maximal treadmill test
  VO2peak is used to describe the cardiorespiratory fitness of the participants
Bone mineral density (BMD) | BMD of the lumbar spine and proximal femur is measured at baseline
  BMD is used to describe the bone health status of the participants
Fat mass (FM) | FM is measured at baseline
  FM is used to describe the body composition of participants
Fat-free mass (FFM) | FFM is measured at baseline
  FFM is used to describe the body composition of participants

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M Kohrt, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Because some journals now require authors to provide access to data, de-identified, anonymized data sets (individual- and group-level data) will be created after study results are published, and made available upon requests for general research purposes, based on availability of resources. To the extent possible, care will be taken to ensure that individual-level data are at very low risk of re-identification and there will be no links to personally identifiable information.
Time Frame: There is no formal plan to share these documents, although requests will be considered. Information related to the protocol and statistical analysis plan will be in the public domain when study results are published.
Access Criteria: Data will become available after publication of study results and be available at least 3 years beyond the completion of the study.

DOCUMENTS (1):
  • Informed Consent Form (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT05029128/ICF_000.pdf